CLINICAL TRIAL: NCT03585478
Title: A Double-Blind, Placebo Controlled, Gluten Challenge Trial of the Efficacy, Safety and Tolerability of 6-weeks Treatment of Latiglutenase (IMGX003) Administration in Patients With Well-Controlled Celiac Disease
Brief Title: Latiglutenase as a Treatment for Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immunogenics, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMGX003-NCCIH-1721; 1R33AT009637-01 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-09

CONDITIONS: Celiac Disease
Keywords: Celiac
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Latiglutenase (Active Comparator): IMGX003
  Interventions: Drug: Latiglutenase
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Latiglutenase — Latiglutenase administered orally (daily)
  Other Names: IMGX003
  Arms: Latiglutenase
Other: Placebo — Placebo administered orally (daily)
  Arms: Placebo

SUMMARY:
Single Center, Randomized, Double-Blind, Placebo Controlled, Gluten Challenge Trial in Patients with Well-Controlled Celiac Disease

DETAILED DESCRIPTION:
This is a phase 2, single-center, prospective, randomized, double-blind, placebo-controlled, study in patients with well-controlled celiac disease. Patients with confirmed CD diagnosis (biopsy) will be recruited to participate in the study. Informed consent must be obtained prior to performing any screening procedures. Patients who meet Visit 1 protocol enrollment criteria will be enrolled and begin the screening period. Patients that fail to meet screening period eligibility will be discontinued from study participation at Visit 2. At Visit 2, eligibility will be confirmed, adverse events will be documented at Visit 2. Patients who continue to meet eligibility requirements at Visit 3 will begin the next treatment phase. During the treatment phase patients will self-administer treatment and gluten daily with their evening meal. At the end of the treatment period, Visit 4, patient eligibility will be confirmed and adverse events will be documented. The final visit, Visit 5, will be a safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed CD diagnosis
* Self-reported adherence to a gluten-free diet for ≥ 12 months
* Agree to maintain dosing of approved prescribed and OTC medications
* Willing to take study treatment with evening meal during any single day
* Willing to take gluten foodstuff with evening meal during any single day
* Willing to maintain GFD for entire study duration
* Willing to agree to minimal ingestion outside of three main daily meals
* Willing and able to comply with all study procedures
* Access to the internet via smartphone, tablet, computer or equivalent to facilitate daily symptom reporting
* Must sign informed consent

Exclusion Criteria:

* Active dermatitis herpetiformis at the time of screening
* IBS (Irritable Bowel Syndrome)
* History of any form of colitis
* Received any systemic biologics (such as monoclonal antibodies or other protein therapeutics where the half-life overlaps with the study start) within 6 months prior to study start
* Taking any oral probiotic supplements (not including probiotics contained in commercially available food preparations) 6 months prior to entry
* Use of any immunosuppressive medications (i.e., for chronic treatment of autoimmune disease or transplant-rejection prophylaxis) 6 months prior to entry
* History of alcohol abuse, illegal drug use
* Unwilling to practice highly effective birth control (unless surgically sterilized or post-menopausal)
* Received any experimental drug within 30 days of randomization, in the case of experimental biologics at least 6 months prior to randomization
* Uncontrolled complications of celiac disease, which, in the opinion of the investigator, could affect immune response or pose an increased risk to the patient
* Inability to give informed consent
* Any medical condition, other than celiac disease, which, in the opinion of the investigator, could adversely affect the patient's participation in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Histologic Protection | 6 weeks
  The primary efficacy endpoint of this study is histologic protection as measured by EGD (Vh:Cd), such that PBO>Latiglutenase

SECONDARY OUTCOMES:
Symptom Severity | 6 weeks
  Mean percent worsening in severity for patient selected GI symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Murray, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - 200 First Street SW, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray JA, Syage JA, Wu TT, Dickason MA, Ramos AG, Van Dyke C, Horwath I, Lavin PT, Maki M, Hujoel I, Papadakis KA, Bledsoe AC, Khosla C, Sealey-Voyksner JA; CeliacShield Study Group. Latiglutenase Protects the Mucosa and Attenuates Symptom Severity in Patients With Celiac Disease Exposed to a Gluten Challenge. Gastroenterology. 2022 Dec;163(6):1510-1521.e6. doi: 10.1053/j.gastro.2022.07.071. Epub 2022 Aug 2. PMID 35931103